CLINICAL TRIAL: NCT03298802
Title: Postpartum Management of Hypertension in Pregnancy With Hydrochlorothiazide: a Randomized Clinical Trial
Brief Title: Postpartum Management of Hypertension in Pregnancy With Hydrochlorothiazide
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 16-0280
Record Dates: First submitted 2017-09-20; First posted 2017-10-02 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Pre-Eclampsia; Gestational Hypertension; Superimposed Pre-Eclampsia; Hypertension, Pregnancy-Induced; Postpartum Pregnancy-Induced Hypertension; Postpartum Preeclampsia
Keywords: readmission; triage visit for pregnancy related hypertension; hydrochlorothiazide
MeSH Terms: conditions — Pre-Eclampsia; Hypertension, Pregnancy-Induced | interventions — Hydrochlorothiazide; Tablets; Sugars

STUDY DESIGN:
Intervention Model Description: double-blind randomized placebo controlled clinical trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: Randomization will be performed by a person not involved in the clinical trial using a computer random list of numbers generated using STATA (StataCorp 14.0, Dallas, TX). This list of random number assignments will be kept secure and sent directly to the investigational drug service (IDS), who will be responsible for the allocation and dispensing of the medications
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Hydrochlorothiazide 50mg Tablet (Active Comparator): Hydrochlorothiazide 50 mg per os once daily as soon as the subjects can tolerate sips of water after delivery and for a total of fourteen days postpartum.
  Interventions: Drug: Hydrochlorothiazide 50mg Tablet
- Placebo Tablet (Placebo Comparator): Placebo per os once daily as soon as the subjects can tolerate sips of water after delivery and for fourteen days postpartum
  Interventions: Drug: Placebo Tablet

INTERVENTIONS:
Drug: Hydrochlorothiazide 50mg Tablet — Hydrochlorothiazide 50 mg per os once daily as soon as the subjects can tolerate sips of water after delivery and for a total of fourteen days postpartum.
  Other Names: HydroDIURIL, Microzide, Esidrix, Oretic
  Arms: Hydrochlorothiazide 50mg Tablet
Drug: Placebo Tablet — Placebo per os once daily as soon as the subjects can tolerate sips of water after delivery and for a total of fourteen days postpartum
  Other Names: sugar pill
  Arms: Placebo Tablet

SUMMARY:
Postpartum prophylactic HCTZ administration for prevention and relapse of preeclampsia or gestational hypertension.

DETAILED DESCRIPTION:
To evaluate effectiveness of hydrochlorothiazide prophylaxis on prophylaxis, prevention and relapse of preeclampsia or gestational hypertension on readmission rates, need for additional antihypertensive therapy and number of triage visits.

ELIGIBILITY:
Inclusion Criteria:

* Maternal age ≥ 18 years and <50 years.
* Diagnosis of gestational hypertension* or preeclampsia^ at any time during pregnancy, labor or postpartum.

  * defined as isolated systolic BP of 140 mm Hg or greater, a diastolic BP of 90 mm Hg or greater, or both) or ^ defines as new-onset hypertension plus new-onset proteinuria, or in the absence of proteinuria, preeclampsia is diagnosed as hypertension in association with thrombocytopenia (platelet count less than 100,000/microliter), impaired liver function (elevated blood levels of liver transaminases to twice the normal concentration), the new development of renal insufficiency (elevated serum creatinine greater than 1.1 mg/dL or a doubling of serum creatinine in the absence of other renal disease), pulmonary edema, or new-onset cerebral or visual disturbances.)

Exclusion Criteria:

* Subject requiring antihypertensive therapy at time of screening.
* Planned discharge with oral anti-hypertensive medication.
* Contraindication to hydrochlorothiazide (advanced renal failure or anuria, hypersensitivity to sulfonamides).
* Subject not able to follow up postpartum.
* Lactose intolerance.
* Pre-gestational diabetes.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women after delivery of neonate
Enrollment: 612 (Estimated)
Dates: Start 2017-11-21 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Rate of readmission and/or triage visits | 1-6 weeks postpartum
  Any visit in the hospital
Need for additional antihypertensive therapy | 1-6 weeks postpartum
  Requiring additional antihypertensive agents in the postpartum period

SECONDARY OUTCOMES:
Length of hospital stay | 1-6 weeks postpartum
  Days that patient required to be in-house in the postpartum period
Total Additional doses of anti-hypertensive therapy | 1-6 weeks postpartum
  Addition of total doses that patient received in the postpartum period
Elevation of blood pressure >150/90 | 1-6 weeks postpartum
  Hypertension definition in the postpartum period
Severe composite maternal morbidity | 1-6 weeks postpartum
  o Any of the following: ICU admission, HELLP syndrome, eclampsia, stroke, renal failure, pulmonary edema, cardiomyopathy or maternal death
Use of resources | 1-6 weeks postpartum
  hospital stay, postpartum clinic or emergency room visit within 4-6 weeks of delivery, need for imaging or other invasive procedures.
Adverse Events | 1-6 weeks Postpartum
  Allergic reactions (anaphylaxis, angioedema, skin rashes including Stevens Johnson and Toxic Epidermal necrolysis)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Bush, M.D., Principal Investigator — UTMB
Locations (2):
- United States (2):
  - St. David's North Austin Medical Center, Austin, Texas
  - University of Texas Medical Branch, Galveston, Texas

IPD SHARING:
Plan to Share IPD: No